CLINICAL TRIAL: NCT03647189
Title: Randomized, Controlled Trial With Hybrid Fractional Laser for Vulvovaginal Atrophy in Breast Cancer Survivors and Menopausal Females
Brief Title: Randomized, Controlled Trial With Hybrid Fractional Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sciton (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIVA-001
Record Dates: First submitted 2018-08-23; First posted 2018-08-27 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Vaginal Atrophy, Sexual Dysfunction, Vaginal Dryness, Dyspareunia
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Dyspareunia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment Arm (Experimental): Subjects will be treated with hybrid fractional laser
  Interventions: Device: Hybrid Fractional Laser
- Control Arm (Placebo Comparator)
  Interventions: Device: Hybrid Fractional Laser

INTERVENTIONS:
Device: Hybrid Fractional Laser — Hybrid Fractional Laser

SUMMARY:
This randomized, controlled trial will evaluate hybrid fractional laser treatment for vulvovaginal atrophy in breast cancer survivors and menopausal females

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy biological female aged between 40 to 70 years 2. Is post-menopausal with a AND b OR c:

  1. No menses for at least 12 months
  2. Follicle-stimulating hormone (FSH) level over 40mlU/mL
  3. Has had a bilateral oophorectomy at least 12 months ago with no hormone replacement 3. Is experiencing at least two self-reported symptoms of GSM, such as

  <!-- -->

  1. Vaginal irritation in the absence of infection
  2. Chronic burning sensation
  3. Chronic itching in the absence of infection
  4. Recurring urinary tract infections (UTIs)
  5. Vaginal dryness during sexual activity
  6. Pain during sexual activity (dyspareunia) 4. Has been experiencing symptoms of GSM for greater than 3 months 5. Is unable due to a medical contraindication or unwilling to receive hormone-based vaginal therapy 6. Early menopause after breast cancer 7. Normal and up to date pap smear, if applicable 8. Is sexually active (i.e. intravaginal intercourse) or has the potential and desire to be sexually active if symptoms of GSM improve 9. Can read, understand and sign informed consent form 10. Has indicated willingness to participate in the study by signing an informed consent form 11. Agrees to adhere to the treatment and follow-up schedule and post treatment care instructions

Exclusion Criteria:

* 1. Undiagnosed abnormal genital bleeding 2. Has history of pelvic surgery or other energy-based vaginal therapy within 12 months prior to enrollment 3. Previous use of topical estrogen therapy within the last 6 months 4. Has used vaginal creams, moisturizers, lubricants or homeopathic preparations, or received anticoagulants, antiplatelet, thrombolytic, vitamin E or anti-inflammatory within 2 weeks of treatment 5. Has history of heart failure 6. Has equal to or greater than stage III prolapse, according to pelvic organ prolapse quantification system (POP-Q) 7. Has an active sexually transmitted infection (STI) 8. Has signs or symptoms of vulvitis/vaginitis 9. Has signs or symptoms of acute urinary tract infection (UTI) 10. Has participated in any clinical trial involving an investigational drug or procedure within past 30 days 11. The investigator feels that for any reason the subject is not eligible to participate in the study

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 25 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Vaginal health index score (VHIS) | 6 months
  Scores vaginal health by scoring it from 1(none) - 5(excellent).
Change from baseline in Female sexual function index questionnaire (FSFI) | 6 months
  Scoring 0(minimum) - 5(maximum)
Change from baseline in day-to-day impact of vaginal aging questionnaire | 6 months
  Questionnaire
Change from baseline in histology | 3 months
  Histology

SECONDARY OUTCOMES:
Change from baseline in photography | 6 months
  Photography

CONTACTS AND LOCATIONS:
Locations (1):
- Miamim Dermatology, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No